CLINICAL TRIAL: NCT05119205
Title: Study of Survival Outcomes of Multiple Myeloma Patients Admitted on Assiut Clinical Hematology Unit Observational Study
Brief Title: Survival Outcomes of Multiple Myeloma Patients Admitted on Assiut Clinical Hematology Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Badr, Assiut University, Assiut University
Other Study IDs: assiut5000
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma Survival Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone marrow biopsy and compete blood count — Bone marrow biopsy and compete blood count will be done for follow up in patients with multiple myeloma

SUMMARY:
Our study will discuss survival outcomes of multiple myeloma patients admitted on Assiut clinical Hematology and role of neutrophil to lymphocyte and lymphocyte to monocyte ratios as prognostic factors in multiple myeloma.

DETAILED DESCRIPTION:
What are survival outcomes and the prognostic value of neutrophil to lymphocyte ratio of multiple myeloma patients admitted on Assiut clinical Hematology unit? Multiple myeloma (MM)is a plasma cell neoplasm associated with its characteristic clinical complications: anemia, infections, renal impairment or bone destruction. MM is the second most commonly diagnosed hematological neoplasm, with an incidence rate of 6.2 per 100 000 individuals .

Survival outcomes have remained constant over the past few decades; therefore, MM is still considered incurable. However, the increasing use of autologous stem cell transplantation (SCT) and the introduction of novel therapeutic agents, such as thalidomide and bortezomib, have improved the survival of myeloma patients .

Relationship between inflammation and cancer have been established. Some inflammatory factors from accessory cells in tumor milieu, such as interleukin-1 (IL-1), IL-6, and tumor necrosis factor-alpha (TNF-α), facilitated cancer cells' invasiveness .

Further studies exhibited the reactive oxygen and nitrogen from inflammatory cells induced mutation of some tumor suppressor genes, and inflammatory factors such as IL-6 and prostaglandin E2 (PGE2) caused DNA methylation, which both played an important role in tumorigenesis. Accordingly, neutrophil to lymphocyte ratio (NLR) coinciding with rationales supported by numerous studies, could offer a precise potency in predicting prognosis of cancers. In fact, many studies already demonstrated the prognostic significance of NLR in various cancers Consistently, a number of meta-analyses further confirmed this view in colorectal cancer, lung cancer, ovarian cancer, breast cancer, and lymphoma and others.

ELIGIBILITY:
Inclusion Criteria: clinical and laboratory diagnosis of multiple myeloma

* multiple myeloma patients received chemotherapy in our unit.

Exclusion Criteria:

* Waldenstrom macroglobulinemia
* MGUS
* Amyloidosis
* Other plasna cell disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with multiple myeloma in our unit will be included in the study and follow-up will be done to determine the outcome.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Determine the survival outcomes of multiple myeloma patients admitted on Assiut clinical Hematology unit | 2 years
  Survival time will be measured as time from index date (that is, diagnosis date for MM patients) to the date of death; patients without a date of death were assumed alive at the end of the study period. Survival estimates will be assessed by types of treatment among MM patients. In addition, the proportion of patients who died or survived at least 2, 3 or 5 years after diagnosis will be also described.

IPD SHARING:
Plan to Share IPD: Undecided